CLINICAL TRIAL: NCT06408740
Title: The Effect of Physical Activity Level on Social Participation, Functioning and Quality of Life in Psychosis Patients
Brief Title: Physical Activity Level in Psychosis Patients
Status: Completed | Type: Observational
Sponsor: Bandırma Onyedi Eylül University (Other)
Responsible Party: Principal Investigator, Hazel Çelik Güzel, PhD, Bandırma Onyedi Eylül University
Other Study IDs: 2023-129
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Psychosis
Keywords: Psychosis; Social Participation; Functioning; Quality of Life; Physical Activity
MeSH Terms: conditions — Psychotic Disorders; Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study was to examine the effect of physical activity level on social participation, functioning and quality of life in patients with psychosis.

DETAILED DESCRIPTION:
Positive and negative symptoms of schizophrenia will be assessed using the Positive and Negative Syndrome Scale, depression will be assessed using the Calgary Depression in Schizophrenia Scale, medication side effects will be assessed using the Glasgow Antipsychotic Side Effect Rating Scale, physical activity level will be assessed using the International Physical Activity Form, social participation will be assessed using the Social Participation Questionnaire, functioning will be assessed using the Brief Functioning Assessment Scale and quality of life will be assessed using the Nottingham Health Profile. The assessments are planned to last 30 minutes for each participant. Participants will be assessed only once and will not be reassessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with schizophrenia and other psychotic disorders according to DSM-V criteria (brief psychosis disorder, schizophreniform disorder, schizoaffective disorder, other disorder with psychosis within the scope of another defined schizophrenia and other disorders with psychosis, other disorders with psychosis within the scope of undefined schizophrenia and other disorders with psychosis), who have had their first episode, who are receiving outpatient treatment
* Whose duration of illness is longer than 2 years
* Being between the ages of 18-65
* Being literate

Exclusion Criteria:

* The participant is in a period of active illness that makes it difficult to conduct research (Positive and Negative Syndrome Scale>70 scale points, Calgary Depression in Schizophrenia Scale score >11 scale points)
* Comorbid psychiatric illness
* The patient has an acute or chronic physical illness that impairs the general medical condition and a disease that will affect cognitive functions (neurological, neoplastic, endocrine and immune disorders, infection, epilepsy or any neurological disease, etc.).
* The patient has a physical illness (loss of limbs, paralysis, etc.) that requires additional care and causes significant disability
* Alcohol and substance use disorder

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only female
Study Population: Psychosis patients
Sampling Method: Non-Probability Sample
Enrollment: 157 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-04-20 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale | 6 months
  The scale is a 30-item semi-structured interview scale with a seven-point severity rating. In our study, individuals scoring below 70 points were included to confirm that the participants were not in the active disease period.
Calgary Schizophrenia Depression Scale | 6 months
  The scale is an interviewer-rated scale and consists of 9 items in four-point Likert type. The cut-off score for schizophrenia accompanied by depressive disorder was determined as 11/12. In our study, individuals scoring below 11 points were included to confirm that the participants were not in a depressive episode.
Glasgow Antipsychotic Side Effect Rating Scale | 6 months
  It is a 22-item self-report scale about the side effects of antipsychotics. An increase in the scale score indicates an increase in the severity of side effects
International Physical Activity Form | 6 months
  This form consists of seven questions and provides information on sitting, walking, moderately vigorous activities and time spent in vigorous activities. The calculation of the total score of the short form includes the sum of duration (minutes) and frequency (days) of walking, moderately vigorous activity and vigorous activity. The sitting score (sedentary behavior level) is calculated separately. Physical activity levels are classified as physically inactive/inactive (<600 MET-min/week), physically inactive/minimally active (600-3000 MET-min/week) and physically active/very active (>3000 MET-min/week).
Community Participation Survey | 6 months
  It is a method used to observe an individual's participation in the community. It consists of 15 headings. It is used to assess individuals' home, family life, social activities and work activities. Home activity is 10 points; social activity is 12 points and work activity is 7 points. The total score from 0 to 29 is calculated.
Brief Functioning Assessment Scale | 6 months
  This scale, which will be used by the researchers, consists of questions designed to measure the extent to which patients experienced difficulties in autonomy, occupational functioning, cognitive functioning, financial issues, interpersonal relations, and leisure time activities during the study. The 24-item scale allows the measurement of 6 different domains of specific functioning: autonomy, occupational, cognitive, financial, interpersonal and leisure activities. The scale provides a total score as well as scores specific to sub-functioning domains. Items are scored according to their severity on a scale of 0 to 4. (0) = no difficulty, (1) = mild difficulty, (2) = moderate difficulty, (3) = severe difficulty. Scores on the scale can range from 0 to 72. A total score above 11 indicates a significant loss of functioning.
Nottingham Health Profile | 6 months
  It is used to assess the quality of life of individuals. It consists of 2 parts. The first part includes six categories of energy, pain, physical mobility, sleep, emotional reactions and social isolation and consists of 38 different questions with yes or no answers. The second part consists of 7 questions. The questionnaire asks about current complaints. Positive answers to specific areas are used to assess severity or the sum of the six categories can be given as a profile. The total score for each of the 6 sub-parameters is between 0 and 100 and the total score for the total score is between 0 and 600. A high score indicates poor quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Bandırma Onyedi Eylül University, Balıkesir, Turkey (Türkiye)